CLINICAL TRIAL: NCT06356337
Title: Light Exposure Tracker in Alzheimer's Disease.
Brief Title: A Light Exposure Tracker Designed to Improve Circadian Rhythms - Aim 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Mariana Figueiro, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY-22-01199
Record Dates: First submitted 2024-04-04; First posted 2024-04-10 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Light Googles plus reminder text messages (Active Comparator): Participants use green light goggles for one hour each morning for two consecutive weeks and also receive a daily text message reminding them to wear the light goggles
  Interventions: Device: Light goggles; Behavioral: Daily reminder test message
- Light Goggles alone (Experimental): Participants use green light goggles for one hour each morning for two consecutive weeks
  Interventions: Device: Light goggles

INTERVENTIONS:
Device: Light goggles — Green light goggles worn for 1 hour each morning for two weeks
Behavioral: Daily reminder test message — Participants will receive daily text message reminding them to use light goggles each morning
  Arms: Light Googles plus reminder text messages

SUMMARY:
The purpose of this research study is to investigate the relationship between reminder messages sent via text and compliance with a daily morning light intervention designed to advance the circadian clock. Twenty healthy adults will be recruited to participate in a randomized, cross-over study where daily messages are, or are not, provided to remind participants to carry out the intervention.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults over the age of 55
* score of 25 or greater on MoCA

Exclusion Criteria:

* Severe sleep apnea
* restless leg syndrome
* obstructing cataracts
* macular degeneration
* diabetic retinopathy
* glaucoma
* use of sleep medications
* brain disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-22 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
Saliva samples for melatonin levels | Baseline and 2-weeks post-intervention for each Arm
  Serial saliva samples will be collected to calculate dim light melatonin onset.

SECONDARY OUTCOMES:
Light exposure using the Speck | worn all 12 study weeks
  The Speck light meter will be used to collect overall light exposure.The Speck light meter uses a photosensor to measure the amount of light study participants are exposed to each day.
Sleep time using actigraphy | worn all 12 study weeks
  Sleep time will be calculated from the actigraph. The wrist actigraph measures activity during the day and how well you sleep at night. The actigraph software will calculate the amount of time spent in bed sleeping.

CONTACTS AND LOCATIONS:
Overall Officials: Mariana Figueiro, PhD, Principal Investigator — Ichan School of Medicine
Locations (1):
- Light and Health Research Center, Menands, New York, United States

IPD SHARING:
Plan to Share IPD: No
overall study results will be shared not individual.